CLINICAL TRIAL: NCT05318547
Title: Assessing Women's Preferences for Postpartum Thromboprophylaxis: the PREFER-PostPartum
Acronym: PREFER-PP
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fondation Hôpital Saint-Joseph (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: PREFER-PP
Record Dates: First submitted 2021-12-30; First posted 2022-04-08 (Actual); Last update posted 2023-08-09 (Actual); Status verified 2023-08

CONDITIONS: Pregnancy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- standard-gamble technique (Experimental): Participants will be asked to imagine a scenario in which they are experiencing one of the 4 described conditions in the long-term. They will declare their preference between (a) keeping this long-term condition as is, or using a painless hypothetical cure that is associated with some risk of death, with the help of a visual aid on a laptop or tablet. A ping-pong technique will be applied until the point of equipoise is reached, when there is indecision whether to take the treatment or not. The utility will be calculated as 1 - the obtained risk of death of the point of equipoise. Health states will be evaluted in different orders across participants.
  The elicitation of health state utilites by the standard-gamble technique is further clarified.
  Interventions: Other: standard-gamble technique
- time trade-off technique (Experimental): Participants will be asked to declare their preference between 50 years of life with the symptoms of 1 of the conditions, or 50-X years without these symptoms, with the help of a visual aid on a laptop or tablet. A ping-pong technique will be applied until the point of equipoise is reached, when there is indecision on the preference of the 2 choices. The utility will be calculated as the 50-x/50 obtained at this point of equipoise. Health states will be evaluted in different orders across participants.
  Interventions: Other: time trade-off technique

INTERVENTIONS:
Other: standard-gamble technique — Participants will be asked to imagine a scenario in which they are experiencing one of the 4 described conditions in the long-term. They will declare their preference between (a) keeping this long-term condition as is, or using a painless hypothetical cure that is associated with some risk of death, with the help of a visual aid on a laptop or tablet. A ping-pong technique will be applied until the point of equipoise is reached, when there is indecision whether to take the treatment or not. The utility will be calculated as 1 - the obtained risk of death of the point of equipoise. Health states will be evaluted in different orders across participants.
  The elicitation of health state utilites by the standard-gamble technique is further clarified.
  Arms: standard-gamble technique
Other: time trade-off technique — Participants will be asked to declare their preference between 50 years of life with the symptoms of 1 of the conditions, or 50-X years without these symptoms, with the help of a visual aid on a laptop or tablet. A ping-pong technique will be applied until the point of equipoise is reached, when there is indecision on the preference of the 2 choices. The utility will be calculated as the 50-x/50 obtained at this point of equipoise. Health states will be evaluted in different orders across participants.
  Arms: time trade-off technique

SUMMARY:
The risk of venous thromboembolism (VTE), which consists of deep vein thrombosis (DVT) and pulmonary embolism (PE), increases during pregnancy and most strikingly in the postpartum period (6 weeks after delivery). Extensive research efforts have led to the identification of many risk factors for VTE events. Examples of such factors include maternal characteristics (personal history of VTE, thrombophilia, obesity, race) and obstetrical characteristics (methods of delivery, pre-term delivery, growth retardation). These allow care providers to risk stratify women at the time of delivery into low, moderate and high-risk women, based on experts' opinion. Further, a risk score, which was recently developed and validated on English and Swedish populations, estimates the risk of postpartum VTE in individuals.

Thromboprophylaxis (TPX) focuses on the use of short-term low-molecular-weight heparin (LMWH). LMWH is believed to reduce the risk of VTE by 50-70%, but the evidence is indirect, with a lack of large-scale randomized trial in the setting of the postpartum period. Further, LMWH is both inconvenient (subcutaneous injections) and possibly associated with haemorrhagic side effects. Alternative drugs do not exist, because direct oral anticoagulants (DOAC) and aspirin are not studied in this setting and because DOAC are contra-indicated in pregnancy and breastfeeding.

Given the unclear balance of benefits and risks, current guidelines vary greatly in the proportion of women with recommended TPX. Gassmann et al. have recently demonstrated, among a cohort of parturients at the Geneva University Hospitals: a recommendation of postpartum TPX in 40.1% of women, with an estimated mean risk of postpartum VTE of 0.12%, according to the 2015 UK guidelines (RCOG), and a recommendation of postpartum TPX in 8.7% of women, with an estimated mean risk of postpartum VTE of 0.20%, according to the 2018 US guidance (ACOG).These low risks of VTE to trigger a recommendation of TPX use contrast with that of experts' opinions, which advocate for a threshold of VTE risk of 1-3% to recommend the use of TPX. Currently, all women delivering by C-section in Geneva receive TPX regardless of their VTE risk.

This dramatic discrepancy of TPX guidance between guidelines, and between guidelines and individual experts, highlights the uncertainty in this setting. Womens' preferences would be critically important here, to guide a rationale and desired use of TPX. Quite surprisingly, such preferences have never been elicited, in spite of the very large number of births every year (5 and 4 million in Europe and the US, respectively).

To inform prescription patterns of postpartum TPX, investigators propose to conduct this prospective study to elicit values and preferences of pregnant and postpartum women.

ELIGIBILITY:
Inclusion Criteria:

* Women aged ≥18 years
* Ongoing pregnancy or in the early postpartum period (within 7 days of delivery)
* Participants may be with or without prior VTE or major bleeding, and with or without previous/current use of postpartum TPX.
* Fluency in French
* Women are able and willing to give free, informed and written consent

Exclusion Criteria:

* Fetal or neonatal death, in order not to bother women during their mourning.
* Women under tutorship or curatorship
* Women deprived of liberty
* Women under court protection There will be no further exclusion criteria, to maximize the external validity of the study.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Estimated)
Dates: Start 2022-05-13 (Actual); Primary Completion 2024-01-12 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Definition of the Threshold of Risk for Postpartum Venous Thromboembolism | Day 1
  This outcome corresponds to the threshold of risk of postpartum Venous thromboembolism at which women prefer the use of short-term postpartum TPX with LMWH over no treatment.

SECONDARY OUTCOMES:
Correlation of the time of interview (antenatal vs. postnatal) with the risk threshold | Day 1
  This outcome corresponds to the determinants of this threshold within the time of interview (antenatal vs. postnatal).
Correlation of demographic factors with the risk threshold | Day 1
  This outcome corresponds tof this threshold within the time of interview (antenatal vs. postnatal), demographic factors.
Correlation of medical factors with the risk threshold | Day 1
  This outcome corresponds to tDeterminants of this threshold within the time of interview (antenatal vs. postnatal) medical factors.
Correlation of obstetric factors with the risk threshold | Day 1
  This outcome corresponds to the Determinants of this threshold within the time of interview (antenatal vs. postnatal), obstetrical factors.

CONTACTS AND LOCATIONS:
Overall Officials: Justine P Hugon Rodin, MD, Principal Investigator — Fondation Hôpital Saint-Joseph
Locations (1):
- Groupe Hospitalier Paris Saint-Joseph, Paris, France

REFERENCES:
- [Background] Pomp ER, Lenselink AM, Rosendaal FR, Doggen CJ. Pregnancy, the postpartum period and prothrombotic defects: risk of venous thrombosis in the MEGA study. J Thromb Haemost. 2008 Apr;6(4):632-7. doi: 10.1111/j.1538-7836.2008.02921.x. Epub 2008 Jan 31. PMID 18248600
- [Background] Blondon M, Quon BS, Harrington LB, Bounameaux H, Smith NL. Association between newborn birth weight and the risk of postpartum maternal venous thromboembolism: a population-based case-control study. Circulation. 2015 Apr 28;131(17):1471-6; discussion 1476. doi: 10.1161/CIRCULATIONAHA.114.012749. Epub 2015 Mar 5. PMID 25745022
- [Background] Blondon M, Harrington LB, Boehlen F, Robert-Ebadi H, Righini M, Smith NL. Pre-pregnancy BMI, delivery BMI, gestational weight gain and the risk of postpartum venous thrombosis. Thromb Res. 2016 Sep;145:151-6. doi: 10.1016/j.thromres.2016.06.026. Epub 2016 Jun 24. PMID 27421192
- [Background] Sultan AA, West J, Grainge MJ, Riley RD, Tata LJ, Stephansson O, Fleming KM, Nelson-Piercy C, Ludvigsson JF. Development and validation of risk prediction model for venous thromboembolism in postpartum women: multinational cohort study. BMJ. 2016 Dec 5;355:i6253. doi: 10.1136/bmj.i6253. PMID 27919934
- [Background] Mismetti P, Laporte S, Darmon JY, Buchmuller A, Decousus H. Meta-analysis of low molecular weight heparin in the prevention of venous thromboembolism in general surgery. Br J Surg. 2001 Jul;88(7):913-30. doi: 10.1046/j.0007-1323.2001.01800.x. PMID 11442521
- [Background] Alalaf SK, Jawad RK, Muhammad PR, Ali MS, Al Tawil NG. Bemiparin versus enoxaparin as thromboprophylaxis following vaginal and abdominal deliveries: a prospective clinical trial. BMC Pregnancy Childbirth. 2015 Mar 28;15:72. doi: 10.1186/s12884-015-0515-2. PMID 25884460
- [Background] Bates SM, Rajasekhar A, Middeldorp S, McLintock C, Rodger MA, James AH, Vazquez SR, Greer IA, Riva JJ, Bhatt M, Schwab N, Barrett D, LaHaye A, Rochwerg B. American Society of Hematology 2018 guidelines for management of venous thromboembolism: venous thromboembolism in the context of pregnancy. Blood Adv. 2018 Nov 27;2(22):3317-3359. doi: 10.1182/bloodadvances.2018024802. PMID 30482767
- See also: Risks of Venous Thromboembolism After Cesarean Section — https://www.practiceupdate.com/content/risks-of-venous-thromboembolism-after-cesarean-section/40288
- See also: Reducing the Risk of Venous Thromboembolism during Pregnancy and the Puerperium — https://www.rcog.org.uk/globalassets/documents/guidelines/gtg-37a.pdf